CLINICAL TRIAL: NCT05835713
Title: Total Intravenous Anesthesia for Rigid Bronchoscopy - Remimazolam Versus Propofol: a Prospective Randomized Controlled Trial
Brief Title: Total Intravenous Anesthesia for Rigid Bronchoscopy Using Remimazolam
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Identically designed study had been published before enrollment of first participant. Therefore, this study was not started. The IRB was approved the withdrawn of the study.
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Professor, Medical Doctor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC 2023-02-076
Record Dates: First submitted 2023-03-21; First posted 2023-04-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Disease; Tracheal Stenosis; Endobronchial Mass
Keywords: Remimazolam; Rigid bronchoscopy
MeSH Terms: conditions — Respiration Disorders; Tracheal Stenosis | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam besylate (Experimental): Remimazolam group receive total intravenous anesthesia using remimazolam besylate and remifentanil during rigid bronchoscopy. Remimazolam group receive flumazenil during the emergence from anesthesia.
  Interventions: Drug: Remimazolam besylate
- Propofol (Active Comparator): Propofol group receive total intravenous anesthesia using propofol and remifentanil during rigid bronchoscopy.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam besylate — Remimazolam group is induced general anesthesia using remimazolam besylate injection (0.2mg/kg bolus). General anesthesia is maintained using remimazolam infusion at a rate of 1mg/kg/h and remifentanil infusion at a rate of 0.05-0.15 mcg/kg/min. After recovering spontaneous respiration during emergence, remimazolam group receive flumazenil injection (0.5 mg)
  Other Names: Byfavo
  Arms: Remimazolam besylate
Drug: Propofol — Propofol group is induced general anesthesia using propofol injection (2 mg/kg bolus). General anesthesia is maintained using propofol infusion at a rate of 4-8 mg/kg/h and remifentanil infusion at a rate of 0.05-0.15 mcg/kg/min.
  Arms: Propofol

SUMMARY:
Rigid bronchoscopy usually requires deep general anesthesia, but the duration of the procedure is relatively short. Remimazolam, a recently developed anesthetics, showed faster recovery from anesthesia and stable hemodynamics compared to propofol, the most popular anesthetics. However, few studies have investigated the usefulness of remimazolam for rigid bronchoscopy. Therefore, the investigators compared the usefulness of propofol and remimazolam in total intravenous anesthesia for rigid bronchoscopy.

DETAILED DESCRIPTION:
Rigid bronchoscopy usually requires deep general anesthesia, but the duration of the procedure is relatively short. Therefore, anesthesiologists need anesthetics that simultaneously provide hemodynamical stability and faster recovery from anesthesia. Remimazolam showed faster recovery from anesthesia and stable hemodynamic profiles compared to propofol, the most popular anesthetics during general anesthesia. However, few studies have investigated the usefulness of remimazolam during rigid bronchoscopy. In this randomized controlled trial, the investigators want to compare the recovery duration from anesthesia after a rigid bronchoscopy procedure between patients undergoing intravenous anesthesia using remimazolam and propofol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who undergoing rigid bronchoscopy under general anesthesia in Samsung Medical Center, Seoul, South Korea
* American Society of Anesthesiologists physical status I, II, III

Exclusion Criteria:

1. patients who are contraindicated in benzodiazepine (e,g., allergy to the drug or have a history of hypersensitivity reactions)
2. drug or alcohol addiction
3. neuromuscular disease or mental illness
4. metabolic disease
5. emergency surgery
6. body mass index >30 kg/m2 or <18.5 kg/m2
7. patient's refusal
8. patients in shock or coma
9. Patients contraindicated to remimazolam such as acute narrow-angle glaucoma, sleep apnea, severe or acute respiratory failure, galactose intolerance, lactase deficiency, glucose-galactose malabsorption, severe hypersensitivity to dextran 40.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
The duration of emergence after rigid bronchoscopy | From the end of anesthetics infusion to the extubation, an average of 10 minutes
  The time interval between the end of anesthetics infusion and the extubation

SECONDARY OUTCOMES:
The duration of induction before rigid bronchoscopy | From the start of anesthetics infusion to the loss of responsiveness, an average of 5 minutes
  Time interval between the start of anesthetics infusion and loss of responsiveness
Awareness during general anesthesia | From the start of anesthetics infusion to the extubation, an average of 30 minutes
  Whether patient experience awareness during general anesthesia. Awareness during general anesthesia will be assessed with the use of a modified Brice questionnaire. 30 minutes after the arrival at a postanesthesia care unit, a study staff who is blind to the allocation of patients will interview the patient.
Use of vasoactive medication during rigid bronchoscopy | From the start of anesthetics infusion to the extubation, an average of 30 minutes
  Whether vasoactive medication is needed to maintain vital signs within 20% of baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No